CLINICAL TRIAL: NCT00827710
Title: Automated Diabetes Registry Tools to Enhance Patient Self-Management and Provider Performance Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Henry Fischer, MD, Denver Health and Hospital Authority
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: AHRQ 290-2006-000-20; AHRQ Contract 290-2006-000-20
Record Dates: First submitted 2009-01-14; First posted 2009-01-23 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes
Keywords: diabetes; registry; computer; self management
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): patients who received point-of-care report cards and were listed on provider performance report card
  Interventions: Behavioral: point of care patient report cards; Behavioral: Provider performance report card
- 2 (Active Comparator): Patients who received point-of-care diabetes report cards but were not listed on provider performance report card
  Interventions: Behavioral: point of care patient report cards
- 3 (Active Comparator): Patients who did not receive point-of-care report card but who were listed on provider performance report card
  Interventions: Behavioral: Provider performance report card
- 4 (No Intervention): Patients who did not receive point of care report card and who did were not listed on provider performance report card

INTERVENTIONS:
Behavioral: point of care patient report cards — gives patient feedback on performance on glycemic, lipid, and blood pressure control relative to expert recommended goals
  Arms: 1; 2
Behavioral: Provider performance report card — Gives provider feedback on performance on their diabetes panel of patients and includes patient level data
  Arms: 1; 3

SUMMARY:
Can we improve diabetes outcomes through 1) report card mailings to patients 2) point of care distribution of report cards to patients and 3) provider performance feedback with patient level data?

DETAILED DESCRIPTION:
Our federally qualified health care center serves over 7000 diabetic patients, many of whom are uninsured (43%) or on medicaid (18%) or medicare (26%). The population is 54% Latino, 25% Caucasian, and 14% African American. We excluded patients older than 75; those without English or Spanish as a first language; and the homeless. The remaining 5457 patients were randomized to this one-year study which ended January 1, 2009. One-half of the enrolled patients received quarterly mailed report cards on their HgA1c, blood pressure, and lipid performance. They were asked to pick from a list of self-management goals and to see their provider if their last visit was more than 2 months prior to the mailing. In a 2x2 design, our eight clinics were randomized to i) on-site printing of patient report cards or no on-site printing and ii) standard provider performance report cards or enhanced provider report cards. The standard provider report cards included data on provider performance on HgA1c, LDL, and blood pressure compared to other providers. The enhanced provider report card also included a list of up to 10 patients not at HgA1c, LDL, or blood pressure goal. The provider report cards were distributed on a quarterly basis, and the point of care patient report cards were distributed at every clinic visit.

We are analyzing the impact of the intervention on the percent of patients at expert recommended goals for glycemic, lipid, and blood pressure control. We are also performing a qualitative analysis to describe provider and patient attitudes toward the interventions.

ELIGIBILITY:
Inclusion Criteria:

* icd9 code for diabetes
* primary care visit in the past 18 months
* English or Spanish as primary language

Exclusion Criteria:

* age more than 75
* No working address

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5457 (Actual)
Dates: Start 2007-12; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Percent of patients with HgA1c < 7 | january 2009
Percent of patients with LDL < 100 mg/dL | january 2009
Percent of patients with BP < 130/80 | january 2009

SECONDARY OUTCOMES:
Percent of patients with A1c checked in last 6 months | january 2009
Percent of patients with LDL checked in past year | january 2009
Percent of patients with BP checked in past year | january 2009

CONTACTS AND LOCATIONS:
Overall Officials: henry h fischer, md, Principal Investigator — Denver Health and Hospital Authority
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

REFERENCES:
- [Derived] Fischer HH, Eisert SL, Durfee MJ, Moore SL, Steele AW, McCullen K, Anderson K, Penny L, Mackenzie TD. The impact of tailored diabetes registry report cards on measures of disease control: a nested randomized trial. BMC Med Inform Decis Mak. 2011 Feb 17;11:12. doi: 10.1186/1472-6947-11-12. PMID 21329495